CLINICAL TRIAL: NCT03541005
Title: Efficacy and Safety of the Obex® Nutritional Supplement in Overweight and Obese Subjects: Phase III.
Brief Title: Evaluation of Obex® in Overweight and Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OBEX-CAT-2018
Record Dates: First submitted 2018-05-03; First posted 2018-05-30 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Nutritional supplement; Weight loss; waist
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obex (Experimental): a nutritional supplement Obex® 8 g daily by oral route divided into two doses of 4g (between 15 and 20 minutes before lunch and dinner) diluted in water or juice for 6 months. Patients will be recommended to comply with a healthy lifestyle through diet and exercise.
  Interventions: Dietary Supplement: Obex
- Placebo (Placebo Comparator): Placebo 8 g daily by oral route divided into two doses of 4g (between 15 and 20 minutes before lunch and dinner) diluted in water or juice for 6 months. Patients will be recommended to comply with a healthy lifestyle through diet and exercise.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Obex — After concluded the six months of treatment, patients will be follow-up during six months without consumption of Obex
  Arms: Obex
Dietary Supplement: Placebo — After concluded the six months of treatment, patients will be follow-up during six months without consumption of the placebo.
  Arms: Placebo

SUMMARY:
* Obesity is an important and growing worldwide
* Obesity is highly related to the development of metabolic syndrome, diabetes, cardiovascular diseases and cancer
* Diverse adverse events have been reported with the use of antiobesity drugs.
* Several articles describe the beneficial effect of several specific components of the Obex® supplement on weight loss, in the reduction of waist circumference, suppression of appetite, decrease fasting glucose levels, improvement of insulin sensitivity and β cells function.
* Therefore, the administration of Obex in overweight and obese patients could be an excellent strategy to induce weight loss and ameliorate the metabolic disturbances related to obesity and overweight.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill the diagnosis criteria of overweight or obesity (BMI ≥ 25.0 and less than 40).
* Age between 20 and 65 years old.
* Values of fasting glucose < 7.0 mmol / L and at two hours < 11.1 mmol / L during Glucose Tolerance Test (OGTT).
* Written informed consent of participation in the study.

Exclusion Criteria:

* Thyroid dysfunction (hypo or hyperthyroidism).
* Type 1 or type 2 diabetes.
* Prediabetes treated with oral agents.
* Alterations of lipids treated with drugs.
* Medicine consumption of or dietary supplements that influence the reduction of body weight.
* Consumption of steroids or prolonged use of them (last 3 months).
* Treatment with immunosuppressive drugs.
* Chronic diseases (of the hepatic, renal and cardiovascular systems, pancreatitis or some type of malignancy condition) or acute at the time of inclusion.
* Insulin resistance due to diseases such as acromegaly, endogenous hypercortisolism, polycystic ovarian syndrome or hyperprolactinemia.
* History of symptomatic hypoglycaemia.
* History of chronic debilitating diseases, anemia and collagen diseases.
* History or existence psychological illness with eating disorders or toxicity.
* History of alcoholism or drug dependence.
* Inability to comply with the instructions of the investigation.
* Severe infections at the time of inclusion.
* Women of childbearing age who use hormonal contraceptives (oral or injectable).
* Pregnant or breastfeeding.
* Known sensitivity to any of the components of the formulation
* Gynoid fat distribution.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Body Weight. | Six months
  Change in body weight from baseline (0) after six months of treatment (i.e., weight at six month minus weight at baseline 0). Body weight measured in kilograms (k).
Change From Baseline in Waist Circumference at Week 24. | Six months
  Change in waist circumference from baseline after six months of treatment (i.e., waist circumference at six month minus waist circumference at baseline 0). Waist measured in centimeters (cm).
To evaluate the effect of Obex® on fasting glucose levels. | Six months
  The primary outcome is to evaluate the effect of the treatment with Obex® on fasting glucose levels by blood analysis.

SECONDARY OUTCOMES:
To evaluate the effect of Obex® on Body Mass Index (BMI). | Six months
  The BMI will be measured by Quételet index.
To evaluate the effect of Obex® on the waist and hip ratio. | Six months
  Waist and hip ratio will be measured according to the World Health Organisation's data gathering protocol.
To evaluate the effect of Obex® on the waist and height ratio. | Six months
  Waist and height ratio will be measured.
To evaluate the effect of Obex® on arterial blood pressures (BP). | Six months
  The arterial BP will be evaluated by the doctor.
To evaluate the effect of Obex® on fasting insulin levels. | Six months
  The insulin levels will be evaluated by blood analysis.
To evaluate the effect of Obex® on insulin resistance. | Six months
  Homeostasis model assessment-estimated insulin resistance (HOMA-IR), calculated from individual serum measures (fasting insulin x fasting glucose/22.5).
To evaluate the effect of Obex® on insulin sensitivity. | Six months
  The Quicki, Bennett and Raynaud insulin sensitivity indexes will be evaluated by QUICKI = [1/[log I0 + log G0], Bennett index (BEN) = 1/(log I0 x log G0), Raynaud index (RAY) = [40/I0]).
To evaluate the effect of Obex® on β-cell function. | Six months
  Homeostatic model assessment-beta cell (HOMA-β), calculated from individual serum measures (20 x fasting insulin (µU/mL)/fasting glucose (mmol/L)-3.5).
To evaluate the effect of Obex® on cholesterol. | Six months
  The cholesterol, triglyceride, HDL-c and LDL-c levels will be evaluated by blood analysis.
To evaluate the effect of Obex® on hepatic enzymes. | Six months
  The hepatic enzymes (Alanine aminotransferase, Aspartate aminotransferase, gamma-glutamyltransferase, Alkaline Phosphatase) will be evaluated by blood analysis.
To evaluate the effect of Obex® on creatinine and uric acid concentrations. | Six months
  The creatinine and uric acid levels will be evaluated by blood analysis.
To evaluate the effect of Obex® on haemoglobin levels. | Six months
  The haemoglobin levels will be evaluated by blood analysis.
To evaluate the effect of Obex® on Conicity Index (CI) | Six months
  CI will be measured by index.

CONTACTS AND LOCATIONS:
Overall Officials: Roselin Valle Cabrera, BSc., Study Director — National Coordinator Center of Clinical Trials (CENCEC)
Locations (1):
- National Institute of Endocrinology, Havana, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Cabrera-Rode E, Cubas-Duenas I, Acosta JR, Hernandez JC, Gonzalez AIC, Calero TMG, Dominguez YA, Rodriguez JH, Rodriguez ADR, Alvarez Alvarez A, Valdes RE, Espinosa LJ, Belent OT, Benavides ZB, Estevez ES, Rodriguez YA, Del Valle Rodriguez J, Julia SM. Efficacy and safety of Obex(R) in overweight and obese subjects: a randomised, double-blind, placebo-controlled clinical trial. BMC Complement Med Ther. 2023 Feb 20;23(1):58. doi: 10.1186/s12906-023-03847-7. PMID 36804035